CLINICAL TRIAL: NCT03186443
Title: Prevention Effect of Pregabalin on Postherpetic Neuralgia: A Multicenter, Randomized, Double-blind, Controlled Trial
Brief Title: Pregabalin Treatment and Prevention Post-herpetic Neuralgia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: China-Japan Friendship Hospital (Other); Nanjing PLA General Hospital (Other); Air Force Military Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TT-01
Record Dates: First submitted 2017-06-07; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Herpetic Neuralgia
Keywords: herpetic neuralgia; post-herpetic neuralgia; pregabalin
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Pregabalin; Gabapentin

STUDY DESIGN:
Intervention Model Description: control group is to oral gabapentin 0.4 tid； experiment group is to oral pregabalin 300mg q 12h
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- pregabalin (Active Comparator): experiment group: pregabalin 300mg,q12h for 6 months
  Interventions: Drug: Pregabalin
- gabapentin (Experimental): compared to pregabalin effect on herpetic neuralgia
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin was taken 300mg,q 12h for 6 month.
  Other Names: pregabalin tablet
  Arms: pregabalin
Drug: Gabapentin — Gabapentin was taken 0.4, tid for 6 month.
  Other Names: gabapentin tablet
  Arms: gabapentin

SUMMARY:
Pregabalin is effective on herpetic neuralgia, but whether can prevention post-herpetic neuralgia still need to confirm.

DETAILED DESCRIPTION:
Pregabalin has been recommended as the first-line drug for post-herpetic neuralgia (PHN) therapy currently due to its efficacy and safety. However,there was no valuable report at present on the clinical efficacy of pregabalin for acute and subacute herpetic neuralgia (SHN), expect for a smaller study which included 29 outpatients who had acute zoster pain for a period of 7-1 4 days. And it is not clear whether early application of pregabalin can reduce the incidence of PHN.

Therefore, this study was rational designed to evaluate the efficacy and safety of pregabalin in the treatment of herpetic neuralgia，and follow-up to the 8 months, evaluation whether impacting the accidence of PHN.

It is the first time in the international that treating acute herpetic neuralgia (AHN) and SHN with pregabalin as a large sample size clinical trial. The results of this study will be great significance for guiding the clinical medication.

ELIGIBILITY:
Inclusion Criteria:

1. Pain occurs within 90 days of rash onset
2. Numerical rating scale (NRS) greater than 50 mm

Exclusion Criteria:

1. Patient with nervous system disorders which impair completing the pain diaries
2. Patient with history of illicit drug or alcohol abuse within the last 2 years

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2017-10-01 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
the changes of numerical rating scale (NRS) | from the date of start to 8 month
  Pain intensity was rated on an 1 1-point numerical rating scale

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | baseline and 8th month
  quality of life was rated on Brief Pain Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Li Wan, Ph.D.,M.D., Study Director — The Second Affiliated Hospital, Guangzhou Medical University
Locations (1):
- National drug clinical trial fundation, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No